CLINICAL TRIAL: NCT04364022
Title: Efficacy of Pragmatic Same-day Ring COVID-19 Prophylaxis for Adult Individuals Exposed to SARS-CoV-2 in Switzerland: an Open-label Cluster Randomized Trial
Brief Title: Efficacy of Pragmatic Same-day COVID-19 Ring Prophylaxis for Adult Individuals Exposed to SARS-CoV-2 in Switzerland
Acronym: COPEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, Prof. Alexandra Calmy, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCER 2020-00864
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Prevention of COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Lopinavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lopinavir/Ritonavir (Active Comparator)
  Interventions: Drug: Lopinavir/ritonavir
- Active surveillance (No Intervention)

INTERVENTIONS:
Drug: Lopinavir/ritonavir — 2x 200mg/50mg, twice daily for 5 days (bid, PO)
  Arms: Lopinavir/Ritonavir

SUMMARY:
A study to assess, in a two-arm open-label cluster randomized clinical trial, the efficacy of a 5-day course of LPV/r treatment in preventing COVID-19 in asymptomatic individuals exposed to a SARS-CoV-2 documented index patient, compared to surveillance alone.

ELIGIBILITY:
Inclusion criteria:

1. Documented close contact with a person with either a PCR-confirmed SARS-CoV-2 or a positive rapid SARS-CoV-2 antigen test (as per standard of care).
2. Enrolment of the participant no more than 7 days since last contact with index case;
3. ≥ 16 years of age;
4. Informed consent as documented by signature (including parent's or legal guardian's signature if the participant is between 16 and 18 y.o.).

Exclusion criteria*:

1. Fever (temperature >38.0°C) and/or respiratory symptoms (cough, dyspnea) and/or new anosmia/ageusia;
2. Individuals with previous confirmed SARS-CoV-2 infection, dating within the last six months ;
3. Known impairment of liver function;
4. Known hypersensitivity to the study medications;
5. Use of any medications that are contraindicated with lopinavir/ritonavir using the website www.hiv-druginteractions.org/checker
6. Individuals on boosted protease inhibitor (other than LPV) or boosted elvitegravir as part of an antiretroviral therapy
7. Inability to be followed-up for the trial period
8. Documented vaccination against SARS-CoV-2

   * Where necessary, additional biological and clinical assessment will be performed, based on clinical judgement.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
21-day incidence of COVID-19 in individuals exposed to SARS-CoV- 2 who are asymptomatic at baseline (intent-to-treat (ITT) analysis). | 21-day

SECONDARY OUTCOMES:
21-day incidence of COVID-19 in individuals exposed to SARS-CoV- 2 who are asymptomatic, PCR-confirmed SARS-CoV-2 negative and have negative SARS-CoV-2 serology at baseline (modified ITT) | 21-day
21-day incidence of SARS-CoV-2 infection in individuals exposed to SARS-CoV-2 who are asymptomatic, PCR-confirmed SARS-CoV-2 negative and have negative SARS-CoV-2 serology at baseline (modified ITT) | 21-day
Severity of clinical COVID-19 on a 7-point ordinal scale | 21-day
  (1: not hospitalized, no limitations on activities, 2: not hospitalized, limitation on activities, 3: hospitalized, not requiring supplemental oxygen, 4: hospitalized, requiring supplemental oxygen, 5: hospitalized, on non- invasive mechanical ventilation 6: hospitalized, on invasive mechanical ventilation or ECMO and 7: death)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Calmy, Prof, Principal Investigator — University Hospital, Geneva; Niklaus Labhardt, Prof, Principal Investigator — Universitätsspital Basel
Locations (4):
- Instituto Nacional de Infectiologia Evandro Chagas, Fiocruz, Rio de Janeiro, Brazil
- Switzerland (3):
  - Universitätsspital Basel and SwissTPH, Basel
  - Hôpitaux Universitaires de Genève, Geneva
  - Ospedale Regionale di Lugano, Lugano

REFERENCES:
- [Derived] Labhardt ND, Smit M, Petignat I, Perneger T, Marinosci A, Ustero P, Diniz Ribeiro MP, Ragozzino S, Nicoletti GJ, Fare PB, Andrey DO, Jacquerioz F, Lebowitz D, Agoritsas T, Meyer B, Spechbach H, Salamun J, Guessous I, Chappuis F, Kaiser L, Decosterd LA, Grinsztejn B, Bernasconi E, Cardoso SW, Calmy A, Team FTCS. Post-exposure Lopinavir-Ritonavir Prophylaxis versus Surveillance for Individuals Exposed to SARS-CoV-2: The COPEP Pragmatic Open-Label, Cluster Randomized Trial. EClinicalMedicine. 2021 Dec;42:101188. doi: 10.1016/j.eclinm.2021.101188. Epub 2021 Nov 6. PMID 34778734
- [Derived] Smit M, Marinosci A, Nicoletti GJ, Perneger T, Ragozzino S, Andrey DO, Stoeckle M, Jacquerioz F, Lebowitz D, Agoritsas T, Meyer B, Spechbach H, Salamun J, Back M, Schaubhut C, Fuchs S, Decosterd L, Battegay M, Guessous I, Chappuis F, Kaiser L, Labhardt ND, Calmy A. Efficacy of pragmatic same-day ring prophylaxis for adult individuals exposed to SARS-CoV-2 in Switzerland (COPEP): protocol of an open-label cluster randomised trial. BMJ Open. 2020 Nov 12;10(11):e040110. doi: 10.1136/bmjopen-2020-040110. PMID 33184083